CLINICAL TRIAL: NCT01913340
Title: Neonatal Erythropoietin And Therapeutic Hypothermia Outcomes Study
Brief Title: Neonatal Erythropoietin And Therapeutic Hypothermia Outcomes in Newborn Brain Injury (NEATO)
Acronym: NEATO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Thrasher Research Fund (Other); Seattle Children's Hospital (Other); Arkansas Children's Hospital Research Institute (Other); Washington University School of Medicine (Other); Children's National Research Institute (Other); Stanford University (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P0055603-01
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Hypoxic-ischemic Encephalopathy; Neonatal Encephalopathy; Birth Asphyxia
Keywords: erythropoietin; therapeutic hypothermia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum | interventions — Erythropoietin; Epoetin Alfa; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erythropoietin (Active Comparator): 1000 U/kg/dose x 5 doses
  Interventions: Drug: Erythropoietin
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Erythropoietin — 1000 U/kg/dose IV x 5 doses
  Other Names: Procrit
  Arms: Erythropoietin
Drug: Normal saline — placebo: NS IV x 5 doses
  Arms: Normal saline

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE), a condition of reduced blood and oxygen flow to a baby's brain near the time of birth, may cause death or neurologic disability. Cooling therapy (hypothermia) provides some protection, but about half of affected infants still have a poor outcome. This clinical trial will determine if the drug erythropoietin, given with hypothermia, is safe to use as a treatment that may further reduce the risk of neurologic deficits after HIE.

DETAILED DESCRIPTION:
This phase I/II clinical trial is designed to demonstrate:

1. The feasibility of recruiting, enrolling and following 50 patients with moderate to severe HIE at 5 sites, while meeting specified recruitment and follow-up target goals.
2. The safety of high-dose Epo therapy in neonates with HIE with respect to systemic organ function and general growth parameters.
3. The value of brain MRI/MRS performed at 4-7 days of age as a biomarker of motor function at 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Newborns ≥ 36 weeks gestation, < 23 hours of age at time of consent, must meet all 3 Inclusion Criteria to be eligible for the study:

  1. Perinatal depression = at least one of the following: a) Apgar ≤5 at 10 min or b) required resuscitation (endotracheal or mask ventilation, or chest compressions) at 10 min or c) pH < 7.0 or base deficit ≥15 in cord, arterial, or venous blood obtained at <60 min of age;
  2. Moderate to severe encephalopathy = at least 3 of 6 modified Sarnat criteria present between 1-6 h of birth: a) reduced level of consciousness; b) decreased spontaneous activity; c) hypotonia; d) decreased suck; e) decreased Moro reflex; or f) respiratory distress including periodic breathing or apnea; and
  3. Hypothermia = passive or active cooling begun by 6 hours of age.

Exclusion Criteria:

* Intrauterine growth restriction (BW <1800 g);
* Major congenital malformation; suspected genetic syndrome, metabolic disorder or TORCH infection;
* Head circumference < 2 SD for gestation;
* Infant for whom withdrawal of supportive care is being considered; or
* Anticipated inability to collect primary endpoint at 12 months of age.

Ages: 30 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne W Wu, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (7):
- United States (7):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - UCSF, San Francisco, California
  - Kaiser Permanente, Santa Clara, Santa Clara, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University, St Louis, Missouri
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Wu YW, Bauer LA, Ballard RA, Ferriero DM, Glidden DV, Mayock DE, Chang T, Durand DJ, Song D, Bonifacio SL, Gonzalez FF, Glass HC, Juul SE. Erythropoietin for neuroprotection in neonatal encephalopathy: safety and pharmacokinetics. Pediatrics. 2012 Oct;130(4):683-91. doi: 10.1542/peds.2012-0498. Epub 2012 Sep 24. PMID 23008465
- [Background] Wu YW, Mathur AM, Chang T, McKinstry RC, Mulkey SB, Mayock DE, Van Meurs KP, Rogers EE, Gonzalez FF, Comstock BA, Juul SE, Msall ME, Bonifacio SL, Glass HC, Massaro AN, Dong L, Tan KW, Heagerty PJ, Ballard RA. High-Dose Erythropoietin and Hypothermia for Hypoxic-Ischemic Encephalopathy: A Phase II Trial. Pediatrics. 2016 Jun;137(6):e20160191. doi: 10.1542/peds.2016-0191. Epub 2016 May 2. PMID 27244862
- [Background] Mulkey SB, Ramakrishnaiah RH, McKinstry RC, Chang T, Mathur AM, Mayock DE, Van Meurs KP, Schaefer GB, Luo C, Bai S, Juul SE, Wu YW. Erythropoietin and Brain Magnetic Resonance Imaging Findings in Hypoxic-Ischemic Encephalopathy: Volume of Acute Brain Injury and 1-Year Neurodevelopmental Outcome. J Pediatr. 2017 Jul;186:196-199. doi: 10.1016/j.jpeds.2017.03.053. Epub 2017 Apr 26. PMID 28456387
- [Background] Darrah J, Bartlett D, Maguire TO, Avison WR, Lacaze-Masmonteil T. Have infant gross motor abilities changed in 20 years? A re-evaluation of the Alberta Infant Motor Scale normative values. Dev Med Child Neurol. 2014 Sep;56(9):877-81. doi: 10.1111/dmcn.12452. Epub 2014 Mar 29. PMID 24684556
- [Background] Massaro AN, Wu YW, Bammler TK, Comstock B, Mathur A, McKinstry RC, Chang T, Mayock DE, Mulkey SB, Van Meurs K, Juul S. Plasma Biomarkers of Brain Injury in Neonatal Hypoxic-Ischemic Encephalopathy. J Pediatr. 2018 Mar;194:67-75.e1. doi: 10.1016/j.jpeds.2017.10.060. PMID 29478510
- [Result] Wu YW, Goodman AM, Chang T, Mulkey SB, Gonzalez FF, Mayock DE, Juul SE, Mathur AM, Van Meurs K, McKinstry RC, Redline RW. Placental pathology and neonatal brain MRI in a randomized trial of erythropoietin for hypoxic-ischemic encephalopathy. Pediatr Res. 2020 Apr;87(5):879-884. doi: 10.1038/s41390-019-0493-6. Epub 2019 Jul 1. PMID 31261373
- [Result] Massaro AN, Wu YW, Bammler TK, MacDonald JW, Mathur A, Chang T, Mayock D, Mulkey SB, van Meurs K, Afsharinejad Z, Juul SE. Dried blood spot compared to plasma measurements of blood-based biomarkers of brain injury in neonatal encephalopathy. Pediatr Res. 2019 Apr;85(5):655-661. doi: 10.1038/s41390-019-0298-7. Epub 2019 Jan 19. PMID 30661082

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erythropoietin | Normal Saline
Started | 24 (22 (92%) received all 5 doses, 1 (4%) received 4 doses, and 1 (4%) only received 1 dose.) | 26
Completed | 21 | 20
Not Completed | 3 | 6
Not completed — Death | 2 | 5
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin | Normal Saline | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age (years)
  years | 29.4 (7.2) | 29.7 (6.6) | 29.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 10 | 16 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Maternal Hispanic ethnicity provided
  Participants
    Hispanic or Latino | 5 | 6 | 11
    Not Hispanic or Latino | 19 | 20 | 39
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Maternal race provided
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 7 | 4 | 11
    White | 14 | 18 | 32
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 3 | 4
Gestational age (weeks) [Mean (Standard Deviation); unit: weeks] — Population: missing data in 1 Epo subject
  weeks
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 38.7 (1.9) | 38.7 (1.6) | 38.7 (1.7)
Maternal education [Count of Participants; unit: Participants] — Population: missing data in 3 Epo and 2 placebo subjects
  Participants
    number analyzed (Participants) | 21 | 24 | 45
    High school or less | 10 | 10 | 20
    Some college or university | 5 | 7 | 12
    College graduate, or post-grad | 6 | 7 | 13
Birth weight (g) [Mean (Standard Deviation); unit: grams] | 3556 (618) | 3243 (512) | 3393 (581)
Large for gestational age [Count of Participants; unit: Participants] | 6 | 1 | 7
Severe Sarnat encephalopathy [Count of Participants; unit: Participants] | 5 | 4 | 9
5 minute Apgar [Count of Participants; unit: Participants] — Apgar score is based on a total score of 1 to 10. Apgar scores of 0-3 are critically low. Apgar scores of 4-6 are below normal. Apgar scores of 7-10 are considered normal. Population: missing data in 1 Epo and 1 placebo subject
  Participants
    number analyzed (Participants) | 23 | 25 | 48
    0-3 (critically low) | 11 | 14 | 25
    4-6 (below normal) | 10 | 10 | 20
    7-10 (normal) | 2 | 1 | 3
10 minute Apgar [Count of Participants; unit: Participants] — Apgar score is based on a total score of 1 to 10. Apgar scores of 0-3 are critically low. Apgar scores of 4-6 are below normal. Apgar scores of 7-10 are considered normal. Population: missing data in 3 Epo and 1 placebo subject
  Participants
    number analyzed (Participants) | 21 | 25 | 46
    0-3 | 5 | 7 | 12
    4-6 | 13 | 11 | 24
    7-10 | 3 | 7 | 10
Resuscitation > 10 minutes [Count of Participants; unit: Participants] — required ongoing resuscitation with chest compressions and/or mechanical ventilation at 10 minutes of age
  Participants | 21 | 21 | 42
Chest compressions [Count of Participants; unit: Participants] | 8 | 11 | 19
Lowest pH [Mean (Standard Deviation); unit: pH] — Lowest pH among cord arterial, cord venous, and arterial blood gas samples taken before 60 minutes of age Population: missing data from 4 Epo and 2 placebo subjects
  pH
    number analyzed (Participants) | 20 | 24 | 44
    (all) | 6.9 (0.2) | 7.0 (0.2) | 6.9 (0.2)
aEEG severe abnormal background [Count of Participants; unit: Participants] — Severe aEEG background at baseline, defined as burst suppression, continuous low voltage or inactive flat tracing Population: missing data from 2 Epo and 2 placebo subjects
  Participants
    number analyzed (Participants) | 22 | 24 | 46
    (all) | 7 | 7 | 14
Maternal chorioamnionitis [Count of Participants; unit: Participants] | 4 | 3 | 7
Delivery mode [Count of Participants; unit: Participants]
  Spontaneous vaginal | 5 | 9 | 14
  Vacuum or forceps | 1 | 2 | 3
  Elective cesarean | 1 | 0 | 1
  Emergency cesarean | 17 | 15 | 32
Sentinel event [Count of Participants; unit: Participants] — placental abruption, shoulder dystocia, uterine rupture or prolapsed cord
  Participants | 7 | 7 | 14
Age at randomization (hours) [Mean (Standard Deviation); unit: hours] — Population: missing data from 2 placebo subjects
  hours
    number analyzed (Participants) | 24 | 24 | 48
    (all) | 13.3 (6.1) | 14.6 (6.1) | 13.9 (6.1)
Age at 1st study drug (hours) [Mean (Standard Deviation); unit: hours] | 15.6 (5.7) | 17.2 (6.1) | 16.5 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Markers of Organ Function
Description: The investigators will monitor organ function and adverse events until hospital discharge from the neonatal intensive care unit
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Measure: Number; unit: participants
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 24 | 26
participants
  Liver dysfunction (ALT >100 IU/L) | 10 | 6
  Hypotension (requiring inotrope or vasopressor) | 9 | 12
  Thrombocytopenia (platelet < 100,000 per uL) | 6 | 10
  Persistent pulmonary hypertension | 5 | 4
  Disseminated intravascular coagulation | 3 | 5
  Sepsis (positive blood culture and antibiotics >=7 | 0 | 5
  Renal dysfunction (creatinine > 1.5) | 4 | 5
  Hypertension (requiring anti-hypertensive) | 1 | 0
  Polycythemia (requiring intervention) | 0 | 0
  Death during birth hospitalization | 2 | 5
  Cardiopulmonary collapse within 2 hours of drug | 1 | 0
  Thrombosis of major vessel | 1 | 1
  Unexpected event related to study drug | 0 | 0

2. Secondary Outcome: Alberta Infant Motor Scale (AIMS)
Description: The AIMS consists of 58 items, including 4 positions: prone (21 items), supine (9 items), sitting (12 items), & standing (16 items). Each item is scored as 'observed' or 'not observed'. Total score range is 0-58, scored as percentile ranks after a raw score is obtained and plotted against age at testing, based on validated norms.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 21 | 20
percentile | 53.5 (5.2) | 42.8 (19.3)

3. Other Pre Specified Outcome: Warner Initial Developmental Evaluation (WIDEA)
Description: A 43-item questionnaire developed and standardized to assess the functional domains of self-care, motor function, communication and social cognition in young children. Self care sub-scale score range 17-68. Mobility score range is 9-36. Communication score range is 13-52. Social Cognition score range is 11-44. Total scale range is 50-200. Higher scores mean higher functioning. Lower scores mean lower functioning.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 21 | 20
units on a scale
  Total score (50-200) | 122 (14) | 110 (31)
  Self-care (17-68) | 36.7 (5.1) | 33.8 (7.7)
  Mobility (9-36) | 28.6 (3.8) | 23.8 (8.9)
  Communication (13-52) | 28.2 (5.1) | 25.5 (8.8)
  Social Cognition (11-44) | 28.8 (6.4) | 26.9 (8.9)

4. Post Hoc Outcome: Warner Initial Developmental Evaluation (WIDEA) at 6 Months of Age
Description: A 43-item questionnaire developed and standardized to assess the functional domains of self-care, motor function, communication and social cognition in young children. Self care score range 7-28. Mobility score range is 9-36. Communication score range is 13-52. Social Cognition score range is 11-44. Higher the score means higher functioning. Lower scores means lower functioning.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 21 | 21
units on a scale
  Total score (50-200) | 75.3 (9.1) | 68.8 (10.7)
  Self-care (7-28) | 28.1 (4.2) | 26.1 (4.7)
  Mobility (9-36) | 14.1 (2.7) | 12.4 (2.7)
  Communication (13-52) | 16.4 (3.2) | 15.3 (2.8)
  Social Cognition (11-44) | 16.7 (4.5) | 14.9 (3.2)

5. Post Hoc Outcome: Moderate to Severe Neurodevelopmental Impairment
Description: Moderate to severe neurodevelopmental impairment at 12 months was defined as AIMS less than 5th percentile for age, or WIDEA more than 2 standard deviations below the mean based on normative data from typically developing infants at 12.9 months of age.
Time Frame: 12-months
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 21 | 20
Participants | 2 | 5

6. Post Hoc Outcome: Growth Parameters: Weight
Time Frame: 12-months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 21 | 20
kg | 9.9 (1.4) | 9.7 (1.2)

7. Post Hoc Outcome: Growth Parameters: Height
Time Frame: 12-months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 21 | 20
cm | 74.3 (3.2) | 71.7 (6.2)

8. Post Hoc Outcome: Growth Parameters: Head Circumference
Time Frame: 12-months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 21 | 20
cm | 45.7 (1.6) | 45.5 (2.1)

9. Post Hoc Outcome: Brain Injury, as Determined by Neonatal Brain MRI
Time Frame: neonatal hospitalization
Population: For subjects randomized to Erythropoietin, age at MRI was 5.6 days (SD 2.8) and subjects received 3.7 (SD 0.8) doses before MRI.
  For subjects randomized to placebo (normal saline), age at MRI was 4.9 days (SD 1.4) and subjects received 3.4 (SD 0.8) doses before MRI.
Measure: Number; unit: participants
Arm/Group | Erythropoietin | Normal Saline
Number analyzed (Participants) | 23 | 25
participants
  Global brain injury score: None (0) | 8 | 3
  Global brain injury score: Mild (1-11) | 14 | 11
  Global brain injury score: Moderate (12-31) | 0 | 6
  Global brain injury score: Severe (>=32) | 1 | 5
  Presence of brain injury: Subcortical | 7 | 17
  Presence of brain injury: Cortical | 4 | 9
  Presence of brain injury: White matter | 12 | 15
  Presence of brain injury: Brainstem | 1 | 4
  Presence of brain injury: Cerebellar | 0 | 5
  Presence of brain injury: >=2 regions injured | 7 | 14

ADVERSE EVENTS:
Description: Adverse Events were only monitored for infants. No Adverse Event data were collected for mothers.
Groups:
- Erythropoietin - Infants: Erythropoietin: 1000 U/kg/dose IV x 5 doses
- Normal Saline - Infants: Normal saline: placebo: NS IV x 5 doses
Arm/Group | Erythropoietin - Infants | Normal Saline - Infants
All-Cause Mortality (participants affected / at risk) | 2/24 | 5/26
Serious Adverse Events (participants affected / at risk) | 3/24 | 6/26
Other Adverse Events (participants affected / at risk) | 17/24 | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erythropoietin - Infants (N=24) | Normal Saline - Infants (N=26)
Cardiopulmonary collapse within 2h of drug (General disorders) | 1 | 0
Thrombosis of major vessel (Blood and lymphatic system disorders) | 1 | 1
Unexpected event related to study drug (General disorders) | 0 | 0
Death during birth hospitalization (General disorders) | 2 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erythropoietin - Infants (N=24) | Normal Saline - Infants (N=26)
Liver dysfunction (ALT >100 IU/L) (Hepatobiliary disorders) | 10 | 6
Hypotension (requiring inotrope or vasopressor) (Vascular disorders) | 9 | 12
Thrombocytopenia (platelet < 100,000 per uL) (Blood and lymphatic system disorders) | 6 | 10
Persistent pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 5
Sepsis (positive blood culture and antibiotics >=7) (Infections and infestations) | 0 | 5
Renal dysfunction (creatinine >1.5) (Renal and urinary disorders) | 4 | 5
Hypertension (requiring anti-hypertensive) (Vascular disorders) | 1 | 0
Polycythemia (requiring intervention) (Blood and lymphatic system disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No